CLINICAL TRIAL: NCT03379701
Title: Applications of Nanotechnology and Chemical Sensors for the Detection and Identification of Chronic Sinusitis Subtypes by Respiratory Samples
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: The Technion (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0037-14
Record Dates: First submitted 2017-11-22; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: CRS
Keywords: chronic rhinosinusitis, nasal polyposis
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — An overall of 2-4 liter breath samples will be collected in inert Mylar bags and immediately transferred to sorbent tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- CRSwPolyps with no Eosonophilia: CRS patients with nasal polyposis, and no eosonophilia.
- CRSwPolyps with Eosonopholia: CRS patients with nasal polyposis and eosonophilia.
- CRS without Polyps: Patients with chronic rhinosinusitis and no nasalpolyposis.
- PCD: Patients with Primrary ciliary dyskinesia .
- AFRS: Patients with allergic fungal rhinosinusitis.
- allergic rhinitis: Patients with allergic rhinitis
- Control: Healthy subjects.

SUMMARY:
Professor Hossam Haick from the Technion, developed an electronic nose for diagnosis of diseases via breath samples.

Biomarkers from nose and sinuses and upper respiratory tract can be detected by "electronic nose".

Identification of biomarkers from nose and sinuses and upper respiratory tract can differentiate between the subtypes of CRS (Chronic rhinosinusitis) and may serve as markers for disease (vs controls), of disease activity (predicting aggressive disease course, predicting Malignant vs Benign nasal "polyps", as inverted papillpma or carcinoma; predicting response to therapy (Steroid , Antibiotics, Nasal wash, Surgery).

DETAILED DESCRIPTION:
Professor Hossam Haick from the Technion, developed an electronic nose for diagnosis of diseases via breath samples.

Biomarkers from nose and sinuses and upper respiratory tract can be detected by "electronic nose".

Identification of biomarkers from nose and sinuses and upper respiratory tract can differentiate between the subtypes of CRS (Chronic rhinosinusitis) and may serve as markers for disease (vs controls), of disease activity (predicting aggressive disease course, predicting Malignant vs Benign nasal "polyps", as inverted papillpma or carcinoma; predicting response to therapy (Steroid , Antibiotics, Nasal wash, Surgery).

The aim of this study is to evaluate various CRS diseases with the Electronic Nose trying to better differentiate CRSwPolyps , CRS without Polyps, PCD, AFS, Vasculitis (as Wegener Granulomatosis) and Allergic Rhinitis with CRS.

For that reason samples were taken from patients from different groups of "CRS patients": 1. CRSwPolyps with no Eosonophilia , 2. CRSwPolyps with Eosonopholia, 3. CRS without Polyps, 4. PCD, 5. AFS, 6. allergic rhinitis and 7. Control subjects.

ELIGIBILITY:
Inclusion Criteria:

1. CRS patients that presented in the Rhinologic clinic at the Hillel Yaffe Medical Center. CRS patients that never had FESS - endoscopic sinus surgery.
2. Willing and able to give inform consent

Control subjects:

1. Age and gender match control individuals that do not have CRS or any other condition that is defined as nasal disease. These individuals will be recruited as "Healthy Population Reference" group.
2. Willing and able to give informed consent

Exclusion Criteria:

1. Patients age 18 or less, pregnant women
2. Presence of HIV, hepatitis or any other potentially severe and infectious disease. Patient that had sinus surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CRS patients will be recruited through the Rhinologic clinic at the Hillel Yaffe Medical Center, after signing an informed consent. Healthy individuals that meet the inclusion/ exclusion criterions will be recruited from among the patient's escorts to the clinic or patients coming for other surgeries (unrelated spouse or acquaintance after signing an informed consent.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2014-09-28 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2016-09-27 (Actual)

PRIMARY OUTCOMES:
discrimination between healthy and CRS subtypes based on SNOT 22 questionnaire results | change in score from recruitment and every six month until 3 years after recruitment.
  SNOT 22 score (score 0-110)
Successful discrimination between healthy and CRS subtypes based on sensor response (electrical resistance measurements) | Change of electrical resistance from recruitment and every six month until 3 years after recruitment.
  Electrical resistance-Disease diagnosis based on breath analysis data classification using an artificial olfactory system (AKA, Electronic nose)

IPD SHARING:
Plan to Share IPD: Undecided